CLINICAL TRIAL: NCT06564922
Title: Effects of Individualized Immediate Postnatal Counselling on Exclusive Breast Feeding During First Month at Bule Hora University Teaching Hospital and Yabelo General Hospital, Oromia, Ethiopia
Brief Title: Effects of Individualized Immediate Postnatal Counselling on Exclusive Breast Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bule Hora University (Other)
Responsible Party: Principal Investigator, Belda Negesa Beyene, Principal Investigator, Bule Hora University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: BuleHoraU
Record Dates: First submitted 2024-08-12; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Breast Feeding; Counselling
Keywords: Breast feeding; Early initiation of breast feeding; Exclusive breast feeding; Immediate counselling; Randomized controlled trial; Oromia; Ethiopia
MeSH Terms: conditions — Breast Feeding | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: The study will have two arms, i.e., intervention and control groups. The intervention group will receive immediate postnatal breastfeeding counselling and control group will receive routine care.
Who Masked: Outcomes Assessor
Masking Description: The intervention will be single-blinded. The outcome assessors will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postnatal Counselling on Exclusive Breast Feeding (Experimental): Counseling on exclusive breastfeeding (EBF) emphasizes starting within the first hour after birth and maintaining it for six months. It covers feeding frequency, proper positioning, and attachment techniques to enhance breastfeeding effectiveness. Benefits include reduced neonatal infections and lower maternal disease risks. The counseling warns against mixed feeding, which can lead to increased infection susceptibility and malnutrition. It also highlights postpartum danger signs in newborns, such as fever and irritability, encouraging early medical intervention. This comprehensive approach aims to empower mothers with knowledge, promoting healthier breastfeeding practices and improving outcomes for both mother and child.
  Interventions: Other: Counselling
- Individualized Immediate Postnatal Counselling on Exclusive Breast Feeding (No Intervention): Usual counselling will be given.

INTERVENTIONS:
Other: Counselling — Counselling was given for treatment group.
  Arms: Postnatal Counselling on Exclusive Breast Feeding

SUMMARY:
Breastfeeding is crucial for the health of both mothers and infants, promoting healthier populations and reducing long-term healthcare costs. To maximize these benefits, education, support, and effective policies are essential. This study aimed to evaluate the impact of immediate postpartum counseling on early initiation and exclusive breastfeeding rates in the pastoralist areas of Oromia, Ethiopia.

Hypothesis: Individualized immediate postnatal counselling improve exclusive breastfeeding practice.

DETAILED DESCRIPTION:
Breastfeeding plays a crucial role in promoting the health and well-being of both mothers and their infants, contributing to healthier populations, and reducing long-term healthcare costs. Encouraging breastfeeding through education, support, and policies is essential for maximizing these benefits. This study aimed to evaluate the impact of immediate postpartum counseling on early initiation of breastfeeding rates and exclusive breastfeeding in Bule Hora and Yabelo Hospitals. A cluster randomized single-blinded trial was conducted on 224 pregnant women (112 for the intervention group and 112 for the control group) from January 1, 2023, to April 30, 2023. The effect of immediate postpartum counselling and its associated variables on early initiation and exclusive breastfeeding practices were evaluated using multiple logistic regressions. A p-value of less than 0.05, a 95% confidence interval, and an adjusted odd ratio were used to determine statistical significance.

ELIGIBILITY:
Inclusion Criteria

* Gave birth by spontaneous vaginal delivery
* Residents of either Yabelo or Bule Hora town hospital
* willing to participate in the study Exclusion Criteria
* Seriously ill and planned to move during the study period
* Stillbirth
* Neonatal death
* Gave birth cesarean delivery

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Early initiation of breastfeeding | up to 1month
  Mothers will be asked about their infant breastfeeding practices, specifically regarding the early initiation of breastfeeding. The practice of early infant breastfeeding initiation will be determined using the operational definition of those who started breastfeeding within one hour after birth, while those who did not initiate breastfeeding within the first hour will be categorized accordingly.

SECONDARY OUTCOMES:
Breastfeeding frequency | up to 1 month
  Frequency of breast-feeding: This section describes the practice of mothers feeding their infants breast milk on demand. In this study, instances where mothers fed their babies according to their needs and the program guidelines were coded as "0," while instances where babies required feeding were coded as "1." Therefore, a code of "1" indicates that the mother frequently breastfed, whereas a code of "0" indicates that she did not frequently breastfeed.
Mother knowledge and attitude | up to 1 month
  Knowledge was assessed by evaluating their understanding of the benefits of breastfeeding for both themselves and their newborns. This evaluation involved eight specific questions. Mothers who answered at or above the mean score were classified as knowledgeable, while those who scored below the mean were considered not knowledgeable.
  Attitude: This study assesses attitudes through 10 questions on a five-point likert scale ranging from "strongly agree" to "strongly disagree." Responses are then simplified into a two-point scale (agree or disagree), with "1" assigned for agreement on positive questions and "0" for disagreement. The reverse applies for negative questions. A positive attitude is indicated by responses that meet or exceed the mean score for breastfeeding items, while scores below the mean indicate a negative attitude.

CONTACTS AND LOCATIONS:
Overall Officials: Belda N Beyene, MSc, Principal Investigator — Bule Hora University, Ethiopia
Locations (1):
- Bule Hora and Yabelo Hospital, Bulē, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: No